CLINICAL TRIAL: NCT04892875
Title: A Phase Ib Study of Concurrent Chemoradiation in Combination With or Without PD1 Inhibitor AB122 Adenosine 2a Receptor / Adenosine 2b Receptor Inhibitor AB928 Therapies in Locally Advanced Head and Neck Cancers (PANTHEoN)
Brief Title: A Study of Concurrent Chemoradiation in Combination With or Without PD1 Inhibitor AB122 Adenosine 2a Receptor / Adenosine 2b Receptor Inhibitor AB928 Therapies in Locally Advanced Head and Neck Cancers
Acronym: PANTHEoN
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding
Sponsor: Jennifer Choe (Other)
Collaborators: Arcus Biosciences, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Jennifer Choe, Assistant Professor of Medicine, Vanderbilt-Ingram Cancer Center
Organization: Vanderbilt-Ingram Cancer Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VICC-VCHAN23126P
Record Dates: First submitted 2021-04-27; First posted 2021-05-19 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Head and Neck Cancer; Squamous Cell Carcinoma of Head and Neck; Oral Cavity Squamous Cell Carcinoma; Oral Cavity Cancer; Oropharynx Cancer; Oropharynx Squamous Cell Carcinoma; Larynx Cancer; Pharynx Cancer; Hypopharynx Cancer; Hypopharynx Squamous Cell Carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Mouth Neoplasms; Oropharyngeal Neoplasms; Laryngeal Neoplasms; Pharyngeal Neoplasms; Hypopharyngeal Neoplasms | interventions — zimberelimab; Cisplatin; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Concurrent Cisplatin/Radiation Therapy + Zimberelimab (Cohort 1) (Experimental): Concurrent weekly cisplatin with radiation and zimberelimab therapy followed by adjuvant zimberelimab
  Interventions: Drug: Zimberelimab; Drug: Cisplatin; Radiation: Radiation
- Concurrent Cisplatin/Radiation Therapy + Zimberelimab + Etrumadenant (Cohort 2) (Experimental): Concurrent weekly cisplatin with radiation + etrumadenant + zimberelimab with adjuvant combined etrumadenant + zimberelimab
  Interventions: Drug: Zimberelimab; Drug: Etrumadenant; Drug: Cisplatin; Radiation: Radiation
- Concurrent Cisplatin/Radiation Therapy (Active Comparator): Concurrent weekly cisplatin with radiation therapy control arm
  Interventions: Drug: Cisplatin; Radiation: Radiation

INTERVENTIONS:
Drug: Zimberelimab — Zimberelimab will be administered at a dose of 360 mg IV on Day 1 of each 21-day cycle for up to 11 cycles.
  Other Names: AB122
  Arms: Concurrent Cisplatin/Radiation Therapy + Zimberelimab (Cohort 1); Concurrent Cisplatin/Radiation Therapy + Zimberelimab + Etrumadenant (Cohort 2)
Drug: Etrumadenant — Etrumadenant will be administered at a dose of 150 mg by mouth once daily on days 1-21 of each 21-day cycle for up to 11 cycles.
  Other Names: AB928
  Arms: Concurrent Cisplatin/Radiation Therapy + Zimberelimab + Etrumadenant (Cohort 2)
Drug: Cisplatin — Concurrent weekly cisplatin and radiation will be administered as part of the subject's standard of care. Cisplatin and radiation will be initiated on the same day and continue for up to 7.5 weeks.
Radiation: Radiation — Concurrent weekly cisplatin and radiation will be administered as part of the subject's standard of care. Cisplatin and radiation will be initiated on the same day and continue for up to 7.5 weeks.

SUMMARY:
The purpose of this study is to test the safety and tolerability of chemotherapy and radiation in combination with the investigational study drugs zimberelimab (AB122) and etrumadenant (AB928) in subjects with a locally advances head or neck cancer. The study will also ask how the study drugs change the following:

* The microbiome that lives in the mouth and on the skin
* Immune cells as they respond to a skin wound
* Scarring (fibrosis) caused by radiation

After completing a screening phase, subjects will be assigned to one of three cohorts:

* Cohort 1: Subjects who will receive cisplatin, radiation and zimberelimab followed by zimberelimab only.
* Cohort 2: Subjects who will receive cisplatin, radiation, zimberelimab and etrumadenant followed by zimberelimab and etrumadent.
* Cohort 3: Subjects who will receive cisplatin and radiation followed by an observation period.

All three cohorts will be followed for a 24 months following the conclusion of the chemoradiation.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the criteria below apply.

1. Age ≥ 18 years of age.
2. Ability to understand and the willingness to sign a written informed consent document.
3. ECOG Performance Status 0-2.
4. Histologically confirmed head and neck squamous cell carcinoma of the oropharynx, larynx, hypopharynx, or pharynx.
5. Satisfies eligibility criteria for treatment with concurrent cisplatin with radiation for the definitive treatment of head and neck squamous cell carcinomas. Eligibility criteria are as follows: HPV-negative Stage III-IVB or HPV-positive Stages II-III and select stage I patients as per PI discretion.
6. Adequate organ and marrow function defined as the following:

   1. Neutrophils ≥ 1500/μL (in absence of growth factor support)
   2. Platelets ≥ 100 x 103/μL without transfusion
   3. Hemoglobin ≥ 9.0 g/dL
   4. Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or creatinine clearance ≥ 50 mL/min as determined by Cockcroft-Gault equation
   5. Aspartate aminotransferase (AST) ≤ 2.5 x ULN
   6. Alanine aminotransferase (ALT) ≤ 2.5 x ULN
   7. Direct bilirubin ≤ 1.5 x ULN (except participants with Gilbert's syndrome who must have direct bilirubin ≤ 3 x ULN).
   8. WBC count ≥ 2500/μL
   9. Lymphocyte count ≥ 500/μL
   10. Albumin ≥ 25 g/L (2.5 g/dL)

Exclusion Criteria:

Participants are excluded from the study if any of the criteria below apply.

1. Prior treatment for head and neck squamous cell carcinoma including systemic therapies, local therapies or radiation.
2. Major medical or other conditions that might affect the study assays: major surgery or trauma in the past 28 days, known current pregnancy, poorly controlled diabetes (repeated glucose >250), history of or current clinically relevant coagulation abnormalities, as determined by the PI. Tracheostomy and feeding tube placement are permitted at any time.
3. Known additional malignancy within the past 3 years (exceptions: basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma-in-situ that have undergone curative therapy).
4. Active or documented history of autoimmune disease or history of a syndrome that required disease-modifying agents, systemic steroids (>10 mg prednisone per day or equivalent) or immunosuppressive medications, except for vitiligo, endocrinopathies in participants stable on hormone replacement therapy, or resolved childhood asthma/atopy within the past 2 years. Participants with asthma requiring intermittent use of bronchodilators (such as albuterol) will not be excluded from this study. Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement for adrenal or pituitary insufficiencies) is not considered a form of systemic treatment and is allowed. This exclusion criteria applies only to Cohorts 1 and 2 but would be allowed on to Cohort 3.
5. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection requiring systemic antibiotic therapy, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, or psychiatric illness/social situations that would limit compliance with study requirements in the opinion of the Investigator or PI.
6. History of myocardial infarction within 6 months or history of arterial thromboembolic event within 3 months of the first dose of investigational agent.
7. Known infection with hepatitis B virus, hepatitis C virus or human immunodeficiency virus (HIV).
8. History of idiopathic pulmonary fibrosis, organizing pneumonia (eg, bronchiolitis obliterans), drug induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan.
9. Grade ≥ 3 hemorrhage or bleeding event within 28 days prior to initiation of study treatment.
10. Cohort 2 only: Inability to swallow medications.
11. Cohort 2 only: Malabsorption condition that would alter the absorption of orally administered medications.
12. Evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding (i.e., in the absence of therapeutic anticoagulation); INR or aPTT ≥ 1.5 ULN.
13. Use of medications that are likely to significantly affect wound healing or clotting (e.g. steroids, anti-coagulants, aspirin > 325 mg per day or other NSAID more once per day).
14. Treatment with therapeutic oral or intravenous (IV) antibiotics within 2 weeks prior to initiation of study treatment. Patients receiving prophylactic antibiotics (eg, to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.

    a. Topical antibiotics are not permitted within 24 hours from the collection "Skin biopsy Pair 1" if the areas of application are anticipated to interfere with the anticipated sites of biopsies.
15. Use of systemic steroids >10 mg prednisone (or equivalent) within 7 days prior to the collection of "Skin biopsy Pair 1" with the exception of pulse dose steroids the day prior to and after CT for prevention of a contrast allergy.
16. Use of any live attenuated vaccines against infectious diseases (e.g., influenza, varicella) within 4 weeks (28 days) of initiation of investigational product.
17. Prior treatment with an anti-PD-L1, anti-PD-1, anti-CTLA-4, or other immune checkpoint inhibitor or agonist as monotherapy or in combination.
18. Use of other investigational drugs (drugs not marketed for any indication) within 28 days or at least 5 half-lives (whichever is longer) before investigational product administration.

    In addition, participants are excluded from Cohort 2 if any of the criteria below apply.
19. Prior treatment with an agent targeting the adenosine pathway.
20. Treatment with known breast cancer resistance protein (BCRP) substrates with a narrow therapeutic window, administered orally (eg, prazosin, rosuvastatin) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment.
21. Treatment with known P-glycoprotein (P-gp) substrates with a narrow therapeutic window, administered orally (eg, digoxin) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment
22. Treatment with known strong CYP3A4 inducers (eg, rifampin, phenytoin, carbamazepine, phenobarbital, and St. John's Wort) and strong CYP3A4 inhibitors (eg, clarithromycin, grapefruit juice, itraconazole, ketoconazole, posaconazole, telithromycin, and voriconazole) within 4 weeks or 5 half lives of the drug (whichever is longer) prior to initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12-31 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events, summarized by attribute and grade, as assessed by using NCI CTCAE v5.0. | Through 30 days after the last dose of study drug
  Toxicity data will be summarized by attribute and grade using NCI CTCAE v5.0.
Tolerability of inhibition with concurrent chemoradiation treatment with or without PD1 inhibition and with or without the adenosine 2A receptor (A2AR) and adenosine 2B receptor (A2BR) as measured by incidence of dose limiting toxicities (DLTs). | From first dose of study drug through 4 weeks after the completion of the radiation therapy
  Incidence of dose limiting toxicities (DLTs)
Effect on imaging correlates of inhibition with concurrent chemoradiation treatment with or without PD1 inhibition and with or without the adenosine 2A receptor (A2AR) and adenosine 2B receptor (A2BR) | Baseline and month 3 of adjuvant period
  Correlation between peripheral immune response and radiographic imaging factors.Correlation between peripheral immune response and radiographic imaging factors.
  Radiographic imaging outcomes for radiation fibrosis based on ARFI and SWEI will be correlated to 1) proportion of change in peripheral immune cell populations and 2) tissue specimens from dermal wound assay expression fold changes of stromal and immune infiltrating markers (e.g. PCR, IHC).
Effect on signaling pathways of immune regulation of inhibition with concurrent chemoradiation treatment with or without PD1 inhibition and with or without the adenosine 2A receptor (A2AR) and adenosine 2B receptor (A2BR) | Prior to first dose of study drugs, Cycle 1 Day 1 (Day 1), Cycle 2 Day 1 (Day 22), Cycle 3 Day 8 (Day 55)and Cycle 11 Day 1 (Day 211). Each cycle is 21 days.
  Measurement of plasma biomarker: soluble CD37
Effect on signaling pathways of immune regulation of inhibition with concurrent chemoradiation treatment with or without PD1 inhibition and with or without the adenosine 2A receptor (A2AR) and adenosine 2B receptor (A2BR) | Prior to first dose of study drugs, Cycle 1 Day 1 (Day 1), Cycle 2 Day 1 (Day 22), Cycle 3 Day 8 (Day 55)and Cycle 11 Day 1 (Day 211). Each cycle is 21 days.
  Measurement of plasma biomarker: cytokines
Effect on signaling pathways of immune regulation of inhibition with concurrent chemoradiation treatment with or without PD1 inhibition and with or without the adenosine 2A receptor (A2AR) and adenosine 2B receptor (A2BR) | Prior to first dose of study drugs, Cycle 1 Day 1 (Day 1), Cycle 2 Day 1 (Day 22), Cycle 3 Day 8 (Day 55)and Cycle 11 Day 1 (Day 211). Each cycle is 21 days.
  Measurement of plasma biomarker: chemokines
Effect on signaling pathways of immune regulation of inhibition with concurrent chemoradiation treatment with or without PD1 inhibition and with or without the adenosine 2A receptor (A2AR) and adenosine 2B receptor (A2BR) | Prior to first dose of study drugs, Cycle 1 Day 1 (Day 1), Cycle 2 Day 1 (Day 22), Cycle 3 Day 8 (Day 55)and Cycle 11 Day 1 (Day 211). Each cycle is 21 days.
  Measurement of plasma biomarker: peripheral blood mononuclear cells (PBMCs)
Effect on would healing of inhibition with concurrent chemoradiation treatment with or without PD1 inhibition and with or without the adenosine 2A receptor (A2AR) and adenosine 2B receptor (A2BR) | Prior to first dose of study drugs and Cycle 3 Day 1 (Day 43). Each cycle is 21 days.
  Dermal wound healing assay
Effect on fibrosis of inhibition with concurrent chemoradiation treatment with or without PD1 inhibition and with or without the adenosine 2A receptor (A2AR) and adenosine 2B receptor (A2BR) | Prior to first dose of study drugs, Cycle 7 Day 1 (Day 127) and Cycle 11 Day 1 (Day 211). Each cycle is 21 days.
  Quantitative measurements of skin fibrosis using acoustic radiation force impulse (ARFI) and shear wave elasticity imaging (SWEI)
Effect on the cutaneous microbiome of inhibition with concurrent chemoradiation treatment with or without PD1 inhibition and with or without the adenosine 2A receptor (A2AR) and adenosine 2B receptor (A2BR) | Prior to first dose of study drugs, Cycle 1 Day 1 (Day 1), Cycle 3 Day 1 (Day 43), Cycle 3 Day 8 (Day 55). Each cycle is 21 days.
  Changes in shotgun metagenomics sequence analysis of the cutaneous microbiome
Effect on the oral microbiome of inhibition with concurrent chemoradiation treatment with or without PD1 inhibition and with or without the adenosine 2A receptor (A2AR) and adenosine 2B receptor (A2BR) | Prior to first dose of study drugs, Cycle 2 Day 1 (Day 22), Cycle 3 Day 8 (Day 55), Cycle 7 Day 1 (Day 127) and Cycle 11 Day 1 (Day 211). Each cycle is 21 days.
  Changes in shotgun metagenomics sequence analysis of the oral microbiome

SECONDARY OUTCOMES:
Proportion of subjects who exhibit a response to the study drugs | Up to 24 months after the last dose of chemoradiation.
  Response will be assessed by RECIST 1.1
Median progression-free survival (PFS) | Up to 24 months after the last dose of chemoradiation.
  Progression-free survival will be assessed by RECIST 1.1
Proportion of subjects with locoregional recurrence | 1 and 2 years
Median overall survival | Up to 24 months after the last dose of chemoradiation
2-year overall survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Choe, MD, PhD, Principal Investigator — Vanderbilt-Ingram Cancer Center

IPD SHARING:
Plan to Share IPD: No